CLINICAL TRIAL: NCT05844280
Title: The Role of Blood Flow Restriction Therapy in Postop Rehabilitation of Foot and Ankle Injuries
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study never opened
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael Johnson, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300009735
Record Dates: First submitted 2023-03-02; First posted 2023-05-06 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Fracture of Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): receiving physical therapy with BFR+NMES devices used at sub-therapeutic levels
  Interventions: Procedure: BFR+NMES at sub therapeutic level
- Treatment Group (Experimental): receiving physical therapy with BFR+NMES devices used at settings that are deemed by prior studies to be therapeutic
  Interventions: Procedure: BFR+NMES at therapeutic level

INTERVENTIONS:
Procedure: BFR+NMES at therapeutic level — This group will receive therapy with BFR+NMES devices used at settings that are deemed by prior studies to be therapeutic.
  Arms: Treatment Group
Procedure: BFR+NMES at sub therapeutic level — This means that the BFR tourniquet and the NMES device will be at such low settings as to not create the treatment effect but subject will have the equipments on their thigh during exercise
  Arms: Control Group

SUMMARY:
The purpose of the study is to determine the role of blood flow restriction (BFR) + neuromuscular electrical stimulation (NMES) in improving post-operative physical therapy and recovery after ankle fracture surgery. We expect to see improved muscle strength, less muscle wasting, and improved functional recovery after surgery when making these additions to routine post-operative (postop) physical therapy protocols.

DETAILED DESCRIPTION:
Few studies have examined BFR in patients sustaining operative foot and ankle injuries. Due to the weight bearing limitations and prolonged immobilization following these injuries, patients often experience increased time away from work and delays with return to sport. These factors are responsible for the rapid muscle atrophy that occurs in the immediate post injury period because of immobility and disuse. Recently, blood flow restriction (BFR) therapy has been shown to be effective in improving muscle strength and preventing atrophy when combined with low load resistance training physical therapy programs.7,8 Neuromuscular electrical stimulation (NMES) is an adjunctive agent that has been show to augment the effects of BFR alone.4 The null hypothesis is that a 2 week BFR + NMES + low load resistance training program in patients age >= 18 recovering from foot and ankle surgery will have no effect on short term (2 weeks postop) lower extremity muscle hypertrophy or atrophy, patient pain and satisfaction, or functional recovery after foot and ankle surgery.

ELIGIBILITY:
Inclusion Criteria:

* isolated, closed low-energy rotational ankle fracture without prior surgery or implants to injured area

Exclusion Criteria:

* history of Deep Vein Thrombosis in affected extremity
* history of significant cardiac disease defined as a recent stent placement in past
* history of peripheral arterial disease
* history of sickle cell disease
* history of coagulopathy
* presenting to surgery >14 days after injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-08 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Assess for calf muscle atrophy as measured by calf circumference | 2 weeks postop
  Calf circumference will be measured using a measuring tape
Assess for calf muscle atrophy as measured by hand held dynamometry | 2 weeks postop
  Hand held Dynamometry will be used to measure the length-tension relationship of the muscle in pounds

SECONDARY OUTCOMES:
Patient tolerance of the BFR treatment using the Visual Analogue Pain Scale. | 2 weeks postop
  The Visual Analogue Pain Scale is used during the beginning, midpoint, and end of a session.
  This scale ranges from 0-10 which 0 being "no pain" and 10 being "worst pain"
Patient tolerance of the BFR treatment using the the Borg Rating of Perceived Exertion f | 2 weeks postop
  The Borg Rating of Perceived Exertion will be used for each session and exercise.
  This rating ranges from 6-20 with 6 being no exertion at all, and 20 being maximum effort

IPD SHARING:
Plan to Share IPD: No